CLINICAL TRIAL: NCT01953510
Title: Evaluation of Different Infant Vaccination Schedules Incorporating Pneumococcal Vaccination
Brief Title: Trial of Pneumococcal Vaccine Schedules in Ho Chi Minh City, Vietnam
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Institut Pasteur (Industry); Menzies School of Health Research (Other); National Health and Medical Research Council, Australia (Other); Bill and Melinda Gates Foundation (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 09/19; 566792 (Other Grant/Funding Number: NHMRC Project Grant); 10PN-PD-DIT-079 (Other: GlaxoSmithKline Biologicals)
Record Dates: First submitted 2013-09-25; First posted 2013-10-01 (Estimated); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Pneumococcal Vaccines
Keywords: Pneumococcal vaccines; 10-valent pneumococcal vaccine; 13-valent pneumococcal vaccine; Immunization Schedule; Public Health
MeSH Terms: interventions — 10-valent pneumococcal conjugate vaccine; PHiD-CV vaccine; 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- A: 3+1 PCV10 (Active Comparator): PCV10 administered at 2, 3, 4 and 9 months of age
  Interventions: Biological: PCV10
- B: 3+0 PCV10 (Experimental): PCV10 administered at 2, 3 and 4 months of age
  Interventions: Biological: PCV10
- C: 2+1 PCV10 (Experimental): PCV10 administered at 2, 4 and 9 months of age
  Interventions: Biological: PCV10
- D: 1+1 PCV10 (Experimental): PCV10 administered at 2 and 6 months of age
  Interventions: Biological: PCV10
- E: 2+1 PCV13 (Experimental): PCV13 administered at 2, 4 and 9 months of age
  Interventions: Biological: PCV13
- F: control (No Intervention): No infant PCV vaccination. PCV10 administered at 18 and 24 months of age
- G: control (No Intervention): Recruited at 18 months of age (non-randomised). PCV10 administered at 24 months of age

INTERVENTIONS:
Biological: PCV10 — PCV10 includes serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F and protein D is the main carrier protein
  Other Names: 10-valent pneumococcal conjugate vaccine; Synflorix
  Arms: A: 3+1 PCV10; B: 3+0 PCV10; C: 2+1 PCV10; D: 1+1 PCV10
Biological: PCV13 — PCV13 includes serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F, individually linked to non-toxic diphtheria CRM197 carrier protein
  Other Names: 13-valent pneumococcal conjugate vaccine; Prevenar-13; Prevnar-13
  Arms: E: 2+1 PCV13

SUMMARY:
Pneumococcus is a group of bacteria that can cause pneumonia, meningitis and other diseases. These bacteria normally live in the nose of humans and are spread from person to person by touching or sneezing. There are vaccines available to protect against infection with these bacteria, and pneumococcus is currently the leading vaccine-preventable cause of death in young children. In countries where pneumococcal vaccine (PCV) has been introduced, there has been a big impact on the amount of disease caused by these bacteria. However, many countries, especially developing countries, are yet to introduce PCV as part of their routine immunizations. Currently a total of four doses of PCV is recommended, and the main barrier to vaccine introduction is cost. This study aims to identify a vaccination schedule to make PCV more effective and affordable for Vietnam and other developing countries.

This study has two distinct purposes: 1) to compare different dosage schedules of PCV and 2) to compare different PCV vaccines.

1. Schedules of Synflorix (PCV10) involving a three, two or one dose PCV primary series and two booster options will be compared. Comparisons will be made firstly in terms of measures of immunity to the vaccine, and secondly in terms of the effect of vaccination on the carriage of bacteria in the nose.
2. The responses to PCV10 and Prevenar-13 (PCV13) will be compared, in the schedule most likely to be considered for global use. Again, comparisons will be made in terms of measures of immunity and effect on carriage in the nose.

Infants aged two months will be randomly assigned to one of six study groups and will provide up to four blood samples for analysis of the measures of immunity and five nose swabs for analysis of carriage of bacteria. Infants will be followed up 8-9 times until the age of 24 months. An additional control group will be recruited at 18 months of age and also followed up until 24 months of age.

The results of this study will be used to facilitate decision making, at global and national levels, regarding introduction of PCV.

DETAILED DESCRIPTION:
Introduction

The overall purpose of this study is to investigate simplified childhood vaccination schedules that are more appropriate for developing country use. This study is specifically designed to address two independent questions within a single study:

1. What is the optimal schedule for provision of EPI vaccines with the incorporation of PCV10? Schedules involving a three, two or one dose PCV10 primary series will be evaluated, timed around options for simplification of the Expanded Programme of Immunization (EPI) schedule for developing countries. A simplified schedule with the pneumococcal booster dose brought forward closer to the peak incidence of disease is likely both to increase compliance and vaccine effectiveness. A booster at nine months of age coincides with the usual time for administration of measles vaccine, whereas a booster at six months of age would provide earlier protection and may enable a further abbreviated 1+1 pneumococcal vaccination schedule.
2. How do the responses to PCV vaccination with PCV10 or PCV13 compare? PCV10 and PCV13 are the two PCVs available through the Advanced Market Commitment (AMC) mechanism, a mechanism that provides funds for vaccine introduction into developing countries. However, there have been no studies to date directly comparing these two vaccines. Directly comparing these two vaccines will provide useful information to countries considering introduction of PCV. There are important differences between these vaccines. PCV10 includes ten pneumococcal serotypes and PCV13 includes thirteen. PCV10 uses a non-typeable Haemophilus influenzae (NTHi) Protein D carrier, which may confer protection against H. influenzae, and PCV13 uses a CRM197 carrier. It is of interest to know whether these vaccines differ either in their immunogenicity or their impact on nasopharyngeal (NP) carriage.

Design

Infants will be randomized to one of six study arms (A-F). All infant participants receive four doses of Infanrix-hexa (DTaP-Hib-HBV-IPV) and at least two doses of PCV. The PCV schedules to be evaluated are: a 3+1 PCV10 schedule at 2, 3, 4 and 9 months of age (Arm A); a 3+0 PCV10 schedule at 2, 3 and 4 months of age (Arm B); a 2+1 PCV10 schedule at 2, 4 and 9 months of age (Arm C); a 1+1 PCV10 schedule at 2 and 6 months of age (Arm D); a 2+1 PCV13 schedule at 2, 4 and 9 months of age (Arm E). Arm F, the control group, receives two doses of PCV10 at 18 and 24 months of age. An additional control group (Arm G) will be recruited at 18 months of age and will receive Infanrix-hexa at 18 months of age and a single dose of PCV10 at 24 months of age. Reactogenicity will be assessed following all vaccination visits through the use of diary cards.

Participants from arms A-E will provide six NP swabs for analysis of the NP carriage outcomes, at 2, 6, 9, 12, 18 and 24 months of age; and will provide four blood samples over the course of the trial for analysis of vaccine responses. Blood 1 will be taken four weeks post-primary series; Blood 2 will be taken pre-booster (arms A, C, D and E) or at 9 months of age (subset of arm B); and Blood 3 will be taken four weeks post-booster (arms A, C, D and E) or at 10 months of age (arm B). An additional blood sample will be taken at: 18 months of age for a subset of arms A, B, C, D and E; 2 months of age for a subset of arm A; 6 months of age for a subset of arms B and C; 9 months of age for a subset of arm D; or 3 months of age for a subset of arm E. Participants from the control arms will provide NP swabs at 2, 6, 9, 12, 18 and 24 months of age (arm F) or at 18 and 24 months of age (arm G), and will provide blood samples at 18 (Blood 4), 19 (Blood X) and 24 (Blood Y) months of age.

Objectives

1. What is the optimal schedule for provision of EPI vaccines with the incorporation of PCV10? The primary objective is to compare a 2+1 schedule at 2, 4 and 9 months of age with a 3+1 schedule at 2, 3, 4 and 9 months of age, with a primary outcome of the immunogenicity of PCV10, four weeks post-primary series (Arm C vs. Arm A+B). Secondary objectives are to investigate an experimental 1+1 schedule at 2 and 6 months of age (Arm D vs. Arm A+B and Arm D vs. Arm C), and to assess the impact of a booster dose on carriage (Arm A vs. Arm F and Arm A vs. Arm B).
2. How do the responses to PCV vaccination with PCV10 or PCV13 compare? The primary objective is to compare a PCV13 schedule at 2, 4 and 9 months of age with a PCV10 schedule at 2, 3, 4 and 9 months of age, with a primary outcome of the immunogenicity of PCV, four weeks post-primary series (Arm E vs. Arm A+B). Secondary objectives are to compare a PCV13 schedule at 2, 4 and 9 months of age with a PCV10 schedule at 2, 4 and 9 months of age (Arm E vs. Arm C), and to compare the responses to a single dose of PCV13 or PCV10 (Arm E vs. Arm D).

Other objectives are: to examine the decline in pneumococcal antibody levels over time (Arm B); to describe the serotype profile of transferred maternal pneumococcal antibodies (Arm A); and to describe the early rates of carriage (Arms A-F); to evaluate a single dose of PCV10 at 18 months of age (Arm F); and to evaluate the immunogenicity of Infanrix-hexa at 18 months of age in children who have received three doses of Infanrix-hexa or three doses of Quinvaxem (DTwP-Hib-HBV) in infancy.

Sample Size

The proposed infant sample size is 1200 with an allocation ratio of 3:3:5:4:5:4, resulting in arm sizes of: A=150, B=150, C=250, D=200, E=250, F=200. Sample size calculations were based on the primary outcomes for each of the two study questions: the post-primary series immunogenicity comparing 1) a two dose (Arm C) and three dose (Arm A+B) PCV10 primary series and 2) a two dose PCV13 (Arm E) and three dose PCV10 (Arm A+B) primary series. A non-inferiority margin of 10% difference in absolute risk (Arm A+B minus Arm C or Arm E), as used by regulatory authorities, is deemed clinically significant. The Farrington-Manning (1990) method was used for the sample size/power estimation, assuming one-sided 5% type I error. If the alternative hypotheses of non-inferiority are accepted for at least 7 out of 10 serotypes, overall non-inferiority will be declared. The power for testing individual serotype hypotheses was calculated using PASS Software 2002. The power for rejecting the overall null hypothesis was estimated by simulation, using a tailor-made simulation program written for implementation in Stata with 10,000 replications. A sample size of 1200 results in >99% power for rejecting the overall null hypothesis for each of the two study questions, allowing for 5% loss to follow-up at four weeks post-primary series. An additional 200 participants aged 18 months (Arm G) will be recruited at the same time as participants from Arms A-F reach 18 months of age, bringing the total sample size of the trial to 1400 participants.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 2 months and 2 months plus 2 weeks (Arms A-F) or aged between 18 months and 18 months plus 2 weeks (Arm G)
* No significant maternal or perinatal history
* Born at or after 36 weeks gestation
* Written and signed informed consent from parent/legal guardian
* Lives within approximately 30 minutes of the commune health centre
* Family anticipates living in the study area for the next 22 months (Arms A-F) or 6 months (Arm G)
* Has received three doses of either Infanrix-hexa or Quinvaxem in infancy (Arm G)

Exclusion Criteria:

* Known allergy to any component of the vaccine
* Allergic reaction or anaphylactic reaction to any previous vaccine
* Known immunodeficiency disorder
* Known HIV-infected mother
* Known thrombocytopenia or coagulation disorder
* On immunosuppressive medication
* Administration or planned administration of any immunoglobulin or blood product since birth
* Severe birth defect requiring ongoing medical care
* Chronic or progressive disease
* Seizure disorder
* History of invasive pneumococcal, meningococcal or Haemophilus influenzae type b diseases, or tetanus, measles, pertussis or diphtheria infections
* Receipt of any 2 month vaccines through the EPI program (Arms A-F) or receipt of PCV (Arm G)
* Family plans on giving the infant Quinvaxem or oral polio vaccine (Arms A-F)

Ages: 60 Days to 74 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1400 (Actual)
Dates: Start 2013-09-30 (Actual); Primary Completion 2016-01-27 (Actual); Study Completion 2021-11-08 (Actual)

PRIMARY OUTCOMES:
proportion of children with antibody concentration ≥0.35µg/mL for individual pneumococcal serotypes | 4 weeks post-primary series
  The immunogenicity of PCV will be measured by ELISA in terms of serotype-specific IgG antibody concentrations. Primary comparisons between arms will be made in terms of the proportion of children with antibody concentration ≥0.35µg/mL for the ten serotypes included in both PCVs. An overall conclusion for between arm comparisons will be based on the rejection of at least seven out of the ten individual serotype null hypotheses.

SECONDARY OUTCOMES:
geometric mean concentration (GMC) of pneumococcal serotype-specific IgG | four weeks post-primary series
  measured by ELISA
proportion of children with pneumococcal serotype-specific opsonisation index (OI) ≥8 | four weeks post-primary series
  OIs for selected pneumococcal serotypes will be measured by opsonophagocytic assay (OPA)
proportion of children with four-fold rise in pneumococcal serotype-specific IgG | change from pre-booster to four weeks post-booster
  measured by ELISA
proportion of children with pneumococcal serotype-specific OI ≥8 | four weeks post-booster
  measured by OPA
median number of pneumococcal polysaccharide (PS)-specific memory B cells | four weeks post-booster
  The number of PS-specific memory B cells will be measured by ELISPOT assays.
median proportion of pneumococcal PS-specific memory B cells | four weeks post-booster
  The proportion of PS-specific memory B cells will be measured in relation to the total number of memory B cells.
median number of pneumococcal PS-specific memory B cells | 18 months of age
  measured by ELISPOT
median proportion of pneumococcal PS-specific memory B cells | 18 months of age
  measured by ELISPOT
NP carriage rate of NTHi | 12 months of age
NP carriage rate of vaccine-type (VT) Streptococcus pneumoniae (S. pneumoniae) | 12 months of age
NP carriage rate of non-VT S. pneumoniae | 12 months of age
NP carriage rate of H. influenzae | 12 months of age
Density of NP carriage of S. pneumoniae | 12 months of age
  measured by quantitative real-time PCR (qPCR)
Density of NP carriage of H. influenzae | 12 months of age
  measured by qPCR
NP carriage rate of NTHi | 18 months of age
NP carriage rate of VT S. pneumoniae | 18 months of age
NP carriage rate of non-VT S. pneumoniae | 18 months of age
NP carriage rate of H. influenzae | 18 months of age
NP carriage rate of VT S. pneumoniae | 24 months of age
  assessed primarily by qPCR and microarray

OTHER OUTCOMES:
proportion of children with a measles IgG antibody titre >150mIU/mL | four weeks post-booster
  measured by ELISA
proportion of children achieving protective antibody levels to the components of Infanrix-hexa | four weeks post-primary series
  Protective antibody levels are defined as: >0.1 IU/mL diphtheria IgG, >0.15 IU/mL tetanus IgG, >0.15 µg/mL Hib PRP antigen IgG, and >10 mIU/mL hepatitis B surface antigen IgG.
proportion of children achieving the expected booster-response antibody levels to the components of Infanrix-hexa | four weeks post-booster
  The expected booster-response antibody levels are : >1.0 IU/mL diphtheria IgG, >1.0 IU/mL tetanus IgG, >1.0 µg/mL Hib PRP antigen IgG, and >1000 IU/mL hepatitis B surface antigen IgG.
NP carriage rate of VT S. pneumoniae | 2 months of age
NP carriage rate of non-VT S. pneumoniae | 2 months of age
NP carriage rate of H. influenzae | 2 months of age
NP carriage rate of NTHi | 2 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Edward K Mulholland, MBBS, FRACP, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- Pasteur Institute of Ho Chi Minh City, Ho Chi Minh City, Vietnam

REFERENCES:
- [Derived] Toh ZQ, Ma YY, Temple B, Anderson J, Far HH, Phan TV, Dai VTT, Huu TN, Toan NT, Bright K, Nation ML, Ortika BD, Nguyen C, Smith-Vaughan H, Satzke C, Mulholland K, Licciardi PV. Relationship between IL-17_A and pneumococcal carriage in children aged under two years: data from a randomised controlled trial in Vietnam. Cytokine. 2026 Feb;198:157094. doi: 10.1016/j.cyto.2025.157094. Epub 2025 Dec 23. PMID 41442837
- [Derived] Smith-Vaughan H, Temple B, Trang Dai VT, Hoan PT, Loc Thuy HN, Phan TV, Bright K, Toan NT, Uyen DY, Nguyen CD, Beissbarth J, Ortika BD, Nation ML, Dunne EM, Hinds J, Lai J, Satzke C, Huu TN, Mulholland K. Effect of different schedules of ten-valent pneumococcal conjugate vaccine on pneumococcal carriage in Vietnamese infants: results from a randomised controlled trial. Lancet Reg Health West Pac. 2022 Dec 3;32:100651. doi: 10.1016/j.lanwpc.2022.100651. eCollection 2023 Mar. PMID 36785850
- [Derived] Licciardi PV, Temple B, Dai VTT, Toan NT, Uyen D, Nguyen CD, Phan TV, Bright K, Marimla RA, Balloch A, Huu TN, Mulholland K. Immunogenicity of alternative ten-valent pneumococcal conjugate vaccine schedules in infants in Ho Chi Minh City, Vietnam: results from a single-blind, parallel-group, open-label, randomised, controlled trial. Lancet Infect Dis. 2021 Oct;21(10):1415-1428. doi: 10.1016/S1473-3099(20)30775-1. Epub 2021 Jun 23. PMID 34171233
- [Derived] Temple B, Nation ML, Dai VTT, Beissbarth J, Bright K, Dunne EM, Hinds J, Hoan PT, Lai J, Nguyen CD, Ortika BD, Phan TV, Thuy HNL, Toan NT, Uyen DY, Satzke C, Smith-Vaughan H, Huu TN, Mulholland K. Effect of a 2+1 schedule of ten-valent versus 13-valent pneumococcal conjugate vaccine on pneumococcal carriage: Results from a randomised controlled trial in Vietnam. Vaccine. 2021 Apr 15;39(16):2303-2310. doi: 10.1016/j.vaccine.2021.02.043. Epub 2021 Mar 19. PMID 33745731
- [Derived] Temple B, Toan NT, Dai VTT, Bright K, Licciardi PV, Marimla RA, Nguyen CD, Uyen DY, Balloch A, Huu TN, Mulholland EK. Immunogenicity and reactogenicity of ten-valent versus 13-valent pneumococcal conjugate vaccines among infants in Ho Chi Minh City, Vietnam: a randomised controlled trial. Lancet Infect Dis. 2019 May;19(5):497-509. doi: 10.1016/S1473-3099(18)30734-5. Epub 2019 Apr 8. PMID 30975525
- [Derived] Temple B, Toan NT, Uyen DY, Balloch A, Bright K, Cheung YB, Licciardi P, Nguyen CD, Phuong NTM, Satzke C, Smith-Vaughan H, Vu TQH, Huu TN, Mulholland EK. Evaluation of different infant vaccination schedules incorporating pneumococcal vaccination (The Vietnam Pneumococcal Project): protocol of a randomised controlled trial. BMJ Open. 2018 Jun 8;8(6):e019795. doi: 10.1136/bmjopen-2017-019795. PMID 29884695